CLINICAL TRIAL: NCT04324164
Title: Survival Outcome of EGFR-TKI in Uncommon EGFR Mutant Advanced Non-small Cell Lung Cancer in China
Brief Title: Survival Outcome of EGFR-TKI in Uncommon EGFR Mutant Advanced NSCLC
Status: Recruiting | Type: Observational
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, professor, Hunan Province Tumor Hospital
Other Study IDs: SONICS
Record Dates: First submitted 2020-03-25; First posted 2020-03-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Cohort 1 Uncommon EGFR exon 19del: patients with uncommon EGFR exon 19del
  Interventions: Drug: Third-generation EGFR-TKI
- Cohort 2 EGFR exon 19delins: patients with EGFR exon 19delins
  Interventions: Drug: Third-generation EGFR-TKI
- Cohort 3 EGFR exon 18del: patients with EGFR exon 18del
  Interventions: Drug: EGFR-TKI
- Cohort 4 Common Uncommon Point Mutations: patients with common uncommon point mutations
  Interventions: Drug: EGFR-TKI
- Cohort 5 Rare Uncommon Point Mutations: patients with rare uncommon point mutations
  Interventions: Drug: EGFR-TKI
- Cohort 6 Compound Mutations Uncommon With Uncommon: patients with compound mutations uncommon with uncommon
  Interventions: Drug: EGFR-TKI
- Cohort 7 Compound Mutations Uncommon With Common: patients with compound mutations uncommon with common
  Interventions: Drug: EGFR-TKI

INTERVENTIONS:
Drug: Third-generation EGFR-TKI — Third-generation EGFR-TKI including Osimertinib/Furmonertinib/Almonertinib, etc.
  Groups: Cohort 1 Uncommon EGFR exon 19del; Cohort 2 EGFR exon 19delins
Drug: EGFR-TKI — All EGFR-TKI
  Groups: Cohort 3 EGFR exon 18del; Cohort 4 Common Uncommon Point Mutations; Cohort 5 Rare Uncommon Point Mutations; Cohort 6 Compound Mutations Uncommon With Uncommon; Cohort 7 Compound Mutations Uncommon With Common

SUMMARY:
This study aims to explore Survival Outcome of EGFR-TKI in Uncommon EGFR Mutant Advanced Non-small Cell Lung Cancer in China

DETAILED DESCRIPTION:
inclusion criteria Uncommon EGFR Mutant Advanced Non-small Cell Lung Cancer EGFR G719X, exon 20 insert mutation without any anti-cancer treatment history

ELIGIBILITY:
Inclusion Criteria:

* 18，Advanced Non-squamous Non-small Cell Lung Cancer Confirmed by Histopathology

  * Uncommon EGFR Mutant Advanced NSCLC

Exclusion Criteria:

* Patients with contraindication of chemotherapy
* Pregnant or breast feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Uncommon EGFR Mutant Advanced Non-small Cell Lung Cancer in China
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2020-03-24 (Actual); Primary Completion 2025-12-24 (Estimated); Study Completion 2027-12-24 (Estimated)

PRIMARY OUTCOMES:
PFS | 5 years
  Defined as the time from the beginning of treatment to the first imaging disease progression or death (whichever occurs first)

SECONDARY OUTCOMES:
OS | 5 years
  Defined as the time from the start of treatment to the death of the subject due to any cause.
ORR | 5 years
  Defined as the proportion of subjects achieving a complete remission (CR) or partial remission (PR) among all subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Yongchang Zhang, MD, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Yongchang Zhang, Changsha, Hunan, China